CLINICAL TRIAL: NCT00029484
Title: Tai Chi Chih and Varicella Zoster Immunity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized
Other Study IDs: R21AT000255-01 (NIH)
Record Dates: First submitted 2002-01-11; First posted 2002-01-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

INTERVENTIONS:
Behavioral: Tai chi chih

SUMMARY:
A randomized control trial testing whether a relaxation response based intervention, Tai Chi Chih, will affect Varicella Zoster Virus (VZV) specific immunity measures of psychological adaptation and health function in the older adult.

DETAILED DESCRIPTION:
Both the incidence and severity of Herpes Zoster (HZ) or "Shingles" increase markedly with increasing age, is a painful condition, due to a decline in Varicella Zoster Virus (VZV) specific immunity. Considerable evidence further shows that psychological stresses salient in the older adult correlate with impairments of cellular immunity.

The investigators have observed that Varicella Zoster Immunity is always decreased in individuals with major depression. Moreover, our preliminary data indicates that the presence of depressive symptoms in older adults is associated with a decline of VZV responder cell frequency (VZV-RCF). Taken together, the untoward effects of age and depressive symptoms on VZV immunity raise the question as to whether an alternative medicine intervention might augment VZV specific immunity in the older adult. We have preliminarily shown that administration of a relaxation-response based intervention, Tai Chi Chih (TCC), results in improvements in health functioning and VZV immunity in older adults as compared to controls. TCC is a slow moving meditation comprised of twenty separate standardized movements for use in elderly populations.

This proposed controlled clinical trial aims to: 1) determine whether the practice of TCC for 16 weeks influences Varicella Zoster Virus (VZV) immunity; 2) demonstrate that TCC can produce significant changes in psychological adaptation, health behaviors, and health functioning and well-being; and 3) assess whether changes in psychological adaptation, health behaviors, and health functioning correlate with changes in VZV immunity following TCC in older adults.

We hypothesize that this behavioral intervention that prioritizes treatment of excessive physiological arousal can influence one's affective state with effects on cellular immunity. By standardization of training and practice schedules, TCC offers an important advantage over prior relaxation response based therapies. Focus on older adults at increase risk for HZ and assay of VZV specific cellular immunity has implications for understanding the impact of behavioral factors and an alternative medicine intervention on a clinically relevant endpoint and the ability of the immune system to respond to antigens of infectious pathogens.

ELIGIBILITY:
History of Varicella or long-term resident (greater than or equal to 30 years) in the continental United States.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Irwin MR, Pike JL, Cole JC, Oxman MN. Effects of a behavioral intervention, Tai Chi Chih, on varicella-zoster virus specific immunity and health functioning in older adults. Psychosom Med. 2003 Sep-Oct;65(5):824-30. doi: 10.1097/01.psy.0000088591.86103.8f. PMID 14508027